CLINICAL TRIAL: NCT04188873
Title: Optimized Chronic Care for Smokers: Developing and Implementing Integrated Clinical and Systems Interventions in Primary Care - Cessation Trial
Brief Title: Cessation Screening Project
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0054; 2P01CA180945 (NIH); A534253 (Other: UW Madison); SMPH/MEDICINE/MEDICINE*G (Other: UW Madison); Protocol Version 10/9/2023 (Other: UW Madison)
Record Dates: First submitted 2019-12-04; First posted 2019-12-06 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Intervention Model Description: Daily smokers will be recruited from primary care to participate in a fully crossed, 2x2x2x2 factorial experiment (N=608) that evaluates 4 different factors: 1) Medication Type (Varenicline vs. Combination NRT [C-NRT]), 2) Preparation Medication (4 Weeks vs. Standard), 3) Medication Duration (Extended [24 weeks] vs. Standard [12 weeks]); and 4) Counseling (Intensive vs. Minimal).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (16):
- 12-week Varenicline with Minimal Counseling (Active Comparator): Participants randomized to this intervention will receive one 0.5 mg pill for the first 3 days, starting 1 week prior to the target quit day (TQD). They will then use one 0.5 mg pill twice daily for the next 4 days. After the first week of study medication ramp up, participants will use one 1 mg pill twice daily until 11 weeks post-TQD. Participants randomized to this intervention will receive a brief (15-30 minute) phone or video counseling session 1 week prior to the TQD to promote engagement with free mobile health resources and then a brief (10-20 minute) follow-up phone or video session during the first week post-TQD to mimic a nurse or clinician follow-up after a quit attempt.
  Interventions: Drug: Standard Duration Varenicline; Behavioral: Minimal Counseling
- 12-week Varenicline with 4-Week Preparation Varenicline and Minimal Counseling (Active Comparator): Participants randomized to this intervention will receive one 0.5 mg pill for the first 3 days, starting 4 week prior to the target quit day (TQD). They will then use one 0.5 mg pill twice daily for the next 4 days. After the first week of study medication ramp up, participants will use one 1 mg pill twice daily for the next 3 weeks pre-TQD and until 12 weeks post-TQD. Participants randomized to this intervention will receive a brief (15-30 minute) phone or video counseling session 1 week prior to the TQD to promote engagement with free mobile health resources and then a brief (10-20 minute) follow-up phone or video session during the first week post-TQD to mimic a nurse or clinician follow-up after a quit attempt.
  Interventions: Drug: Preparation Varenicline and Standard Duration Varenicline; Behavioral: Minimal Counseling
- 24-week Varenicline with Minimal Counseling (Active Comparator): Participants randomized to this intervention will receive one 0.5 mg pill for the first 3 days, starting 1 week prior to the target quit day (TQD). They will then use one 0.5 mg pill twice daily for the next 4 days. After the first week of study medication ramp up, participants will use one 1 mg pill twice daily until 23 weeks post-TQD. Participants randomized to this intervention will receive a brief (15-30 minute) phone or video counseling session 1 week prior to the TQD to promote engagement with free mobile health resources and then a brief (10-20 minute) follow-up phone or video session during the first week post-TQD to mimic a nurse or clinician follow-up after a quit attempt.
  Interventions: Drug: Extended Duration Varenicline; Behavioral: Minimal Counseling
- 24-week Varenicline with 4-Week Preparation Varenicline and Minimal Counseling (Active Comparator): Participants randomized to this intervention will receive one 0.5 mg pill for the first 3 days, starting 4 weeks prior to the target quit day (TQD). They will then use one 0.5 mg pill twice daily for the next 4 days. After the first week of study medication ramp up, participants will use one 1 mg pill twice daily for the next 3 weeks pre-TQD and until 24 weeks post-TQD. Participants randomized to this intervention will receive a brief (15-30 minute) phone or video counseling session 1 week prior to the TQD to promote engagement with free mobile health resources and then a brief (10-20 minute) follow-up phone or video session during the first week post-TQD to mimic a nurse or clinician follow-up after a quit attempt.
  Interventions: Drug: Preparation Varenicline and Extended Duration Varenicline; Behavioral: Minimal Counseling
- 12-week Varenicline with Intensive Counseling (Active Comparator): Participants randomized to this intervention will receive one 0.5 mg pill for the first 3 days, starting 1 week prior to the target quit day (TQD). They will then use one 0.5 mg pill twice daily for the next 4 days. After the first week of study medication ramp up, participants will use one 1 mg pill twice daily until 11 weeks post-TQD. Participants randomized to this intervention will receive four 15-20 minute phone or video counseling sessions (1 prior to the TQD, 1 during the first week post-TQD and during Weeks 2 and 4 post-TQD). The counseling is designed to produce intra-treatment support and skill training, consistent with the Public Health Service (PHS) Clinical Practice Guideline.
  Interventions: Drug: Standard Duration Varenicline; Behavioral: Intensive Counseling
- 12-week Varenicline with 4-Week Preparation Varenicline and Intensive Counseling (Active Comparator): Participants randomized to this intervention will receive one 0.5 mg pill for the first 3 days, starting 4 week prior to the target quit day (TQD). They will then use one 0.5 mg pill twice daily for the next 4 days. After the first week of study medication ramp up, participants will use one 1 mg pill twice daily for the next 3 weeks pre-TQD and until 11 weeks post-TQD. Participants randomized to this intervention will receive four 15-20 minute phone or video counseling sessions (1 prior to the TQD, 1 during the first week post-TQD and during Weeks 2 and 4 post-TQD). The counseling is designed to produce intra-treatment support and skill training, consistent with the Public Health Service (PHS) Clinical Practice Guideline.
  Interventions: Drug: Preparation Varenicline and Standard Duration Varenicline; Behavioral: Intensive Counseling
- 24-week Varenicline with Intensive Counseling (Active Comparator): Participants randomized to this intervention will receive one 0.5 mg pill for the first 3 days, starting 1 week prior to the target quit day (TQD). They will then use one 0.5 mg pill twice daily for the next 4 days. After the first week of study medication ramp up, participants will use one 1 mg pill twice daily until 23 weeks post-TQD. Participants randomized to this intervention will receive four 15-20 minute phone or video counseling sessions (1 prior to the TQD, 1 during the first week post-TQD and during Weeks 2 and 4 post-TQD). The counseling is designed to produce intra-treatment support and skill training, consistent with the Public Health Service (PHS) Clinical Practice Guideline.
  Interventions: Drug: Extended Duration Varenicline; Behavioral: Intensive Counseling
- 24-week Varenicline with 4-Week Preparation Varenicline and Intensive Counseling (Active Comparator): Participants randomized to this intervention will receive one 0.5 mg pill for the first 3 days, starting 4 weeks prior to the target quit day (TQD). They will then use one 0.5 mg pill twice daily for the next 4 days. After the first week of study medication ramp up, participants will use one 1 mg pill twice daily for the next 3 weeks pre-TQD and until 24 weeks post-TQD. Participants randomized to this intervention will receive four 15-20 minute phone or video counseling sessions (1 prior to the TQD, 1 during the first week post-TQD and during Weeks 2 and 4 post-TQD). The counseling is designed to produce intra-treatment support and skill training, consistent with the Public Health Service (PHS) Clinical Practice Guideline.
  Interventions: Drug: Preparation Varenicline and Extended Duration Varenicline; Behavioral: Intensive Counseling
- 12-week C-NRT with Minimal Counseling (Active Comparator): Participants randomized to this intervention will receive 12 weeks of nicotine patches and nicotine mini-lozenges to use starting on their quit day. Participants who smoke more than 10 cigarettes/day will start with a 21 mg patch for 8 weeks, and then titrate down to a 14 mg patch for 2 weeks and then a 7 mg patch for 2 weeks. Participants who smoke 5-10 cigarettes/day will be given 10 weeks of 14 mg patches and then 2 weeks of 7 mg patches. Participants will receive 2 mg mini-lozenges. Participants randomized to this intervention will receive a brief (15-30 minute) phone or video counseling session 1 week prior to the TQD to promote engagement with free mobile health resources and then a brief (10-20 minute) follow-up phone or video session during the first week post-TQD to mimic a nurse or clinician follow-up after a quit attempt.
  Interventions: Drug: Standard Duration Combination NRT; Behavioral: Minimal Counseling
- 12-week C-NRT with 4-Week Preparation C-NRT and Minimal Counseling (Active Comparator): Participants randomized to this intervention will receive 14 mg patches starting 4 weeks prior to the target quit day (TQD). Then, starting on the TQD, participants will receive 12 weeks of nicotine patches and nicotine mini-lozenges. Participants who smoke >10 cigarettes/day will start with a 21 mg patch for 8 weeks, and then titrate down to a 14 mg patch for 2 weeks and then a 7 mg patch for 2 weeks. Participants who smoke 5-10 cigarettes/day will be given 10 weeks of 14 mg patches and then 2 weeks of 7 mg patches. Participants will receive 2 mg mini-lozenges. Participants will receive a brief 15-30 minute phone or video counseling session 1 week prior to the TQD to promote engagement with free mobile health resources and then a brief (10-20 minute) follow-up phone or video session during the first week post-TQD to mimic a nurse or clinician follow-up after a quit attempt.
  Interventions: Drug: Preparation Combination NRT and Standard Duration Combination NRT; Behavioral: Minimal Counseling
- 24-week C-NRT with Minimal Counseling (Active Comparator): Participants randomized to this intervention will receive 24 weeks of nicotine patches and nicotine mini-lozenges, starting on the target quit day (TQD). Participants who smoke more than 10 cigarettes/day will start with a 21 mg patch for 20 weeks, and then titrate down to a 14 mg patch for 2 weeks and then a 7 mg patch for 2 weeks. Participants who smoke 5-10 cigarettes/day will be given 22 weeks of 14 mg patches and then 2 weeks of 7 mg patches. Participants will receive 2 mg mini-lozenges. Participants randomized to this intervention will receive a brief (15-30 minute) phone or video counseling session 1 week prior to the TQD to promote engagement with free mobile health resources and then a brief (10-20 minute) follow-up phone or video session during the first week post-TQD to mimic a nurse or clinician follow-up after a quit attempt.
  Interventions: Drug: Extended Duration Combination NRT; Behavioral: Minimal Counseling
- 24-week C-NRT with 4-Week Preparation C-NRT and Minimal Counseling (Active Comparator): Participants randomized to this intervention will receive 14 mg patches starting 4 weeks prior to the target quit day (TQD). Then, starting on the TQD, participants will receive 24 weeks of nicotine patches and nicotine mini-lozenges. Participants who smoke more than 10 cigarettes/day will start with a 21 mg patch for 20 weeks, and then titrate down to a 14 mg patch for 2 weeks and then a 7 mg patch for 2 weeks. Participants who smoke 5-10 cigarettes/day will be given 22 weeks of 14 mg patches and then 2 weeks of 7 mg patches. Participants will receive 2 mg mini-lozenges. Participants will receive a brief (15-30 minute) phone or video counseling session 1 week prior to the TQD to promote engagement with free mobile health resources and then a brief (10-20 minute) follow-up phone or video session during the first week post-TQD to mimic a nurse or clinician follow-up after a quit attempt.
  Interventions: Drug: Preparation Combination NRT and Extended Duration Combination NRT; Behavioral: Minimal Counseling
- 12-week C-NRT with Intensive Counseling (Active Comparator): Participants randomized to this intervention will receive 12 weeks of nicotine patches and nicotine mini-lozenges to use starting on their quit day. Participants who smoke more than 10 cigarettes/day will start with a 21 mg patch for 8 weeks, and then titrate down to a 14 mg patch for 2 weeks and then a 7 mg patch for 2 weeks. Participants who smoke 5-10 cigarettes/day will be given 10 weeks of 14 mg patches and then 2 weeks of 7 mg patches. Participants will receive 2 mg mini-lozenges. Participants randomized to this intervention will receive four 15-20 minute phone or video counseling sessions (1 prior to the TQD, 1 during the first week post-TQD and during Weeks 2 and 4 post-TQD). The counseling is designed to produce intra-treatment support and skill training, consistent with the Public Health Service (PHS) Clinical Practice Guideline.
  Interventions: Drug: Standard Duration Combination NRT; Behavioral: Intensive Counseling
- 12-week C-NRT with 4-Week Preparation C-NRT and Intensive Counseling (Active Comparator): Participants randomized to this intervention will receive 14 mg patches starting 4 weeks prior to the target quit day (TQD). Starting on the TQD, participants will receive 12 weeks of nicotine patches and nicotine mini-lozenges. Participants who smoke >10 cigarettes/day will start with a 21 mg patch for 8 weeks, and then titrate down to a 14 mg patch for 2 weeks and then a 7 mg patch for 2 weeks. Participants who smoke 5-10 cigarettes/day will be given 10 weeks of 14 mg patches and then 2 weeks of 7 mg patches. Participants will receive 2 mg mini-lozenges. Participants will receive four 15-20 minute phone or video counseling sessions (1 prior to the TQD, 1 during the first week post-TQD and during Weeks 2 and 4 post-TQD). The counseling is designed to produce intra-treatment support and skill training, consistent with the Public Health Service (PHS) Clinical Practice Guideline.
  Interventions: Drug: Preparation Combination NRT and Standard Duration Combination NRT; Behavioral: Intensive Counseling
- 24-week C-NRT with Intensive Counseling (Active Comparator): Participants randomized to this intervention will receive 24 weeks of nicotine patches and nicotine mini-lozenges, starting on the target quit day (TQD). Participants who smoke more than 10 cigarettes/day will start with a 21 mg patch for 20 weeks, and then titrate down to a 14 mg patch for 2 weeks and then a 7 mg patch for 2 weeks. Participants who smoke 5-10 cigarettes/day will be given 22 weeks of 14 mg patches and then 2 weeks of 7 mg patches. Participants will receive 2 mg mini-lozenges. Participants randomized to this intervention will receive four 15-20 minute phone or video counseling sessions (1 prior to the TQD, 1 during the first week post-TQD and during Weeks 2 and 4 post-TQD). The counseling is designed to produce intra-treatment support and skill training, consistent with the Public Health Service (PHS) Clinical Practice Guideline.
  Interventions: Drug: Extended Duration Combination NRT; Behavioral: Intensive Counseling
- 24-week C-NRT with 4-Week Preparation C-NRT and Intensive Counseling (Active Comparator): Participants randomized to this intervention will receive 14 mg patches starting 4 weeks prior to the target quit day (TQD). Starting on the TQD, participants will receive 24 weeks of nicotine patches and nicotine mini-lozenges. Participants who smoke >10 cigarettes/day will start with a 21 mg patch for 20 weeks, and then titrate down to a 14 mg patch for 2 weeks and then a 7 mg patch for 2 weeks. Participants who smoke 5-10 cigarettes/day will be given 22 weeks of 14 mg patches and then 2 weeks of 7 mg patches. Participants will receive 2 mg mini-lozenges. Participants will receive four 15-20 minute phone or video counseling sessions (1 prior to the TQD, 1 during the first week post-TQD and during Weeks 2 and 4 post-TQD). The counseling is designed to produce intra-treatment support and skill training, consistent with the Public Health Service (PHS) Clinical Practice Guideline.
  Interventions: Drug: Preparation Combination NRT and Extended Duration Combination NRT; Behavioral: Intensive Counseling

INTERVENTIONS:
Drug: Preparation Varenicline and Standard Duration Varenicline — 16 weeks of varenicline starting 4 weeks pre-quit
  Arms: 12-week Varenicline with 4-Week Preparation Varenicline and Intensive Counseling; 12-week Varenicline with 4-Week Preparation Varenicline and Minimal Counseling
Drug: Preparation Varenicline and Extended Duration Varenicline — 28 weeks of varenicline starting 4 weeks pre-quit
  Arms: 24-week Varenicline with 4-Week Preparation Varenicline and Intensive Counseling; 24-week Varenicline with 4-Week Preparation Varenicline and Minimal Counseling
Drug: Standard Duration Varenicline — 12 weeks of varenicline
  Arms: 12-week Varenicline with Intensive Counseling; 12-week Varenicline with Minimal Counseling
Drug: Extended Duration Varenicline — 24 weeks of varenicline
  Arms: 24-week Varenicline with Intensive Counseling; 24-week Varenicline with Minimal Counseling
Drug: Preparation Combination NRT and Standard Duration Combination NRT — 16 weeks of nicotine patch + nicotine mini-lozenge starting 4 weeks pre-quit
  Arms: 12-week C-NRT with 4-Week Preparation C-NRT and Intensive Counseling; 12-week C-NRT with 4-Week Preparation C-NRT and Minimal Counseling
Drug: Preparation Combination NRT and Extended Duration Combination NRT — 28 weeks of nicotine patch + nicotine mini-lozenge starting 4 weeks pre-quit
  Arms: 24-week C-NRT with 4-Week Preparation C-NRT and Intensive Counseling; 24-week C-NRT with 4-Week Preparation C-NRT and Minimal Counseling
Drug: Standard Duration Combination NRT — 12 weeks of nicotine patch + nicotine mini-lozenge
  Arms: 12-week C-NRT with Intensive Counseling; 12-week C-NRT with Minimal Counseling
Drug: Extended Duration Combination NRT — 24 weeks of nicotine patch + nicotine mini-lozenge
  Arms: 24-week C-NRT with Intensive Counseling; 24-week C-NRT with Minimal Counseling
Behavioral: Intensive Counseling — 4 phone or video counseling sessions
  Arms: 12-week C-NRT with 4-Week Preparation C-NRT and Intensive Counseling; 12-week C-NRT with Intensive Counseling; 12-week Varenicline with 4-Week Preparation Varenicline and Intensive Counseling; 12-week Varenicline with Intensive Counseling; 24-week C-NRT with 4-Week Preparation C-NRT and Intensive Counseling; 24-week C-NRT with Intensive Counseling; 24-week Varenicline with 4-Week Preparation Varenicline and Intensive Counseling; 24-week Varenicline with Intensive Counseling
Behavioral: Minimal Counseling — 2 brief phone or video counseling sessions
  Arms: 12-week C-NRT with 4-Week Preparation C-NRT and Minimal Counseling; 12-week C-NRT with Minimal Counseling; 12-week Varenicline with 4-Week Preparation Varenicline and Minimal Counseling; 12-week Varenicline with Minimal Counseling; 24-week C-NRT with 4-Week Preparation C-NRT and Minimal Counseling; 24-week C-NRT with Minimal Counseling; 24-week Varenicline with 4-Week Preparation Varenicline and Minimal Counseling; 24-week Varenicline with Minimal Counseling

SUMMARY:
This project will use the Multiphase Optimization Strategy (MOST) to guide the development of optimized treatment strategies for the two most effective smoking cessation medications (Combination Nicotine Replacement [C-NRT] and varenicline). The investigators will recruit daily smokers from primary care to participate in a fully crossed, 2x2x2x2 factorial experiment (N=608) that evaluates 4 different factors: 1) Medication Type (Varenicline vs. C-NRT), 2) Preparation Medication (4 Weeks vs. Standard), 3) Medication Duration (Extended [24 weeks] vs. Standard [12 weeks]); and 4) Counseling (Intensive vs. Minimal). Participants will complete assessments one week pre-quit and then assessments of smoking status, treatment use, side effects, potential treatment mechanisms (e.g., withdrawal, self-efficacy) during the first week post-target quit date (TQD) and at Weeks 2, 4, 12, 20, 26, and 52 post-target quit date. These data will be used to examine the main and interactive effects of these four factors on various outcomes, with biochemically confirmed 12-month abstinence serving as the primary outcome. These data will also be used to determine which factors and combinations of factors are most effective with regard to 12-month biochemically confirmed abstinence and cost, thereby identifying optimized varenicline and C-NRT treatments, with each developed to yield especially great benefit. These optimized treatments will then be tested in the Optimized Care Project. The investigators will also examine the relative effects of each medication on particular outcomes (e.g., 12-month abstinence).

DETAILED DESCRIPTION:
Design and Objective: The Cessation Screening Project is a 4-factor factorial screening experiment (i.e., 2x2x2x2 = 16 experimental conditions) designed to identify the most promising intervention components that are especially effective and cost-effective with regard to their main and interactive effects on 12-month biochemically verified abstinence. This design will allow us to: 1) detect main effects and interactions within the factorial experiment and identify especially effective regimens for varenicline and for (Combination Nicotine Replacement) C-NRT; 2) compare the relative effectiveness of varenicline and C-NRT; and 3) identify the most effective and cost-effective counseling intensity to use with the optimized medication regimens. Finally, these results will allow us to identify two optimized treatment packages for use with primary care smokers interested in quitting: packages that include both counseling and pharmacotherapies optimized on the bases of effectiveness and cost.

Recruitment and Participants: Participants (N=608) will be primary care patients from 12 primary care clinics in two Wisconsin healthcare systems. Smokers will be identified via the healthcare system electronic health record (EHR). All EHR-identified smokers in a clinic will receive a mailed invitation to find out more about smoking treatment by calling a healthcare system Care Manager (CM). In addition, using an opt-out strategy, Medical Assistants (MAs), using an EHR-guided prompt, will inform all identified smokers seen at in-person or tele-health visits that they will be contacted by the CM unless the participant indicates s/he wants to opt-out. The participant contact information will then be automatically sent to the CM unless the participant opts out; the investigators have developed and used this workflow successfully in their past research. The CM will call and tell patients about the smoking cessation options available for them including the availability of this smoking cessation study. If patients are interested, the CM will obtain oral assent for screening and sharing contact, primary care team, and screening data with the research team before screening patients for eligibility. Eligible patients will learn more about the study and have a chance to ask questions and provide verbal informed consent. Finally, participants will complete a brief series of questions and then the CM will schedule a call with the study staff (i.e., a Health Counselor) in the database to initiate treatment and complete study assessments. Participants interested in quitting but not eligible for this study will be electronically referred to the Wisconsin Tobacco Quit Line and/or their primary care provider (PCP) by the CM.

Those who agree to and pass the screening for the inclusion/exclusion criteria for study participation will be asked to complete an oral consent and HIPAA authorization process next. After the patient provides oral consent, the CM will notify the patient's PCP via EHR that the patient has volunteered for a study with C-NRT or varenicline. The PCP will notify the CM via the EHR that the patient is medically eligible to receive either agent, as required by the collaborating healthcare systems. This will occur within 5 business days. The PCP will be notified via EHR of the patient's treatment assignment and of study-related serious adverse events or adverse events that prompt medication discontinuation that may occur. Care coordination with the PCP will occur via Tobacco Care Manager entry of data in the patient EHR.

Procedures and Measures: At the second study call, participants (N=608) will be randomized to one level of each of 4 factors: 1) Medication Type (Varenicline vs. C-NRT), 2) Preparation Medication (4 weeks vs. Standard), 3) Medication Duration (Extended vs. Standard), and 4) Counseling (Intensive vs. Minimal). Participants will be told their treatment condition at Call 2, set a target quit date (TQD), and instructed how to use their study medications. Medications will be mailed following this call, along with a handout that describes: 1) when to begin taking study medication; 2) the type and doses involved; 3) how and when to obtain the next month's medication; and 4) complete instructions on proper medication use, including information from the package insert and contact information if they have questions regarding their medication and/or symptoms they experience. Participants will be mailed all Preparation Medication as well as one month of post-quit study medication after Call 2. They will need to call in to a study line to request that more medication be mailed to them (Standard Duration participants will call one time to receive their final 2 months of medication; Extended Duration participants will call once to get 2 additional months of medication and again to get the remaining 3 months of study medication). Participants will also receive a counseling handout with their medications; those randomized to intensive counseling will receive a Quit Plan listing their target quit day and when they start the medications and those randomized to minimal counseling will receive the mobile health (mHealth) handout.

Participants will complete phone assessments one week pre-quit, during the first week post-target quit date (TQD) and at Weeks 2, 4, 12, 20, 26, and 52 post-TQD.

Outcomes: The primary outcome for this study is biochemically confirmed, point-prevalence abstinence at 12 months post-TQD (Primary Aim 1). The secondary outcome is cost effectiveness in which the costs of implementing each intervention (minus research-related costs) will be computed from a payer perspective. Costs will be combined with the intent-to-treat biochemically verified 7-day point prevalence abstinence at 12 months post-TQD to determine the cost per quit.

ELIGIBILITY:
Inclusion Criteria:

* Smoking >4 cigarettes/day for the previous 6 months
* Able to read, write, and speak English
* If currently using nicotine replacement therapy (NRT), agreeing to use only study medication for the duration of the study
* Medically eligible to use study medications
* If the participant is a woman of childbearing potential, using an approved method of birth control during treatment

Exclusion Criteria:

* Currently taking bupropion or varenicline
* Suicidal ideation in the last 12 months or any suicide attempts in the past 10 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 529 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-05-08 (Actual)

PRIMARY OUTCOMES:
Intent-to-treat biochemically verified 7-day point prevalence abstinence | 12 months post-target quit day (TQD)
  Participants will be asked to report on any smoking in the last seven days at a follow-up phone interview scheduled to occur 12-months post-target quit day (post-TQD). Those claiming complete abstinence (not even a puff from a cigarette) in the last seven days at this follow-up interview will be asked to provide a saliva sample for biochemical verification of self-reported abstinence via cotinine testing. Participants who report abstinence in the last 7 days at this visit but have a cotinine level >10ng/mL or who do not have provide a cotinine result will be considered to be smoking.

SECONDARY OUTCOMES:
Cost-effectiveness | 12 months post-target quit day (TQD)
  The costs of implementing each intervention (minus research-related costs) will be computed from a payer perspective. Costs will be combined with the intent-to-treat biochemically verified 7-day point prevalence abstinence at 12 months post-TQD to determine the cost per quit.

CONTACTS AND LOCATIONS:
Overall Officials: Megan E Piper, PhD, Study Director — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - University of Wisconsin Center for Tobacco Research and Intervention, Madison, Wisconsin
  - UW Center for Tobacco Research and Intervention, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
We will make the final de-identified datasets available in standard file formats by request from other researchers in a timely manner (no later than the acceptance for publication of the main findings from the final dataset).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication of the main findings
Access Criteria: Approval of a data request by the investigators

REFERENCES:
- [Derived] Theodoulou A, Chepkin SC, Ye W, Fanshawe TR, Bullen C, Hartmann-Boyce J, Livingstone-Banks J, Hajizadeh A, Lindson N. Different doses, durations and modes of delivery of nicotine replacement therapy for smoking cessation. Cochrane Database Syst Rev. 2023 Jun 19;6(6):CD013308. doi: 10.1002/14651858.CD013308.pub2. PMID 37335995

DOCUMENTS (3):
  • Study Protocol (2023-10-09): https://cdn.clinicaltrials.gov/large-docs/73/NCT04188873/Prot_001.pdf
  • Statistical Analysis Plan (2023-10-09): https://cdn.clinicaltrials.gov/large-docs/73/NCT04188873/SAP_002.pdf
  • Informed Consent Form (2023-08-08): https://cdn.clinicaltrials.gov/large-docs/73/NCT04188873/ICF_000.pdf